CLINICAL TRIAL: NCT05150249
Title: Prospective Observational Study Based on a Cohort of Geriatric Patients With Hip Fracture Treated in the Centers Belonging to the GIOG Group
Acronym: GIOG
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: GIOG
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Hip Fractures; Older Patients; Comprehensive Geriatric Assessment
Keywords: GIOG ( Italian Society of Anesthesiology);; geriatric; orthogeriatric; co-management
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study aims to collect the clinical activity and management data of the Orthogeriatrics and Orthopedics Units participating in the study on a continuous and long-term basis. By collecting clinical data and comparing the performance of the various centers, the study aims to guide the participating centers towards the principles of good clinical practice in orthogeriatrics.

DETAILED DESCRIPTION:
Multicenter prospective cohort observational study. The enrollment period will be 5 years. An additional 4 months will be required to allow the last enrolled patients to complete the 120-day follow-up. It is estimated to enroll a total of 7,000 patients. To facilitate the participation in the study of non-university or IRCCS assistance departments, two methods of data collection will be possible:

* High intensity: continuous data collection for the whole period of the study on all the incident cases
* Low intensity: data collection once a year on incident cases over a continuous period of 1 month, with a reduced number of variables.

The choice of the level of intensity with regard to the data collection method will take place on a voluntary basis (each OU will actually choose the type of speed with which it intends to collaborate in the project, after communicating to the steering committee and to the biostatisticians of the study)

ELIGIBILITY:
Inclusion Criteria:

* Fracture of the femur, regardless of the cause
* Age ≥ 65 years
* Willingness to participate in the study by the patient or a relative / caregiver, if the patient is unable to understand and is not "competent" at the time of the evaluation.
* Able to speak the Italian language

Exclusion Criteria:

* none

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients with a fracture of the femur in which there is a co-management of the clinical problems of the elderly patient between orthopedists and geriatricians
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Estimated)
Dates: Start 2019-07-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Compare the management and clinical methods | Entire study duration, approximately 5 years
  Compare the management and clinical methods of the various centers and evaluate the relationship between indicators of treatment adherence to international guidelines and the short and long-term outcomes of patients.

SECONDARY OUTCOMES:
Circum-annual rhythms of fractures and the multidimensional profiles of patients by age group | Entire study duration, approximately 5 years
  Analyze the circum-annual rhythms of fractures and the multidimensional profiles (clinical, functional and cognitive) of patients by age group
Improvement of clinical practice | Entire study duration, approximately 5 years
  Progressively direct all the centers participating in the study towards the principles of orthogeriatric "good clinical practice", periodically analyzing their performances and comparing them with those established as optimal by the international scientific literature; in this perspective, the study can be configured as a "quality improvement project". In fact, the multidisciplinary discussion and comparison that will follow the systematic review of the indicators analyzed will stimulate, as has already happened elsewhere (e.g. in the United Kingdom), a process of continuous improvement of clinical and surgical practices.
Improvement of collaboration of specialists from various disciplines | Entire study duration, approximately 5 years
  Actively involve specialists from various disciplines who are currently engaged in an uncoordinated way in the management of these patients and seek synergies with other potentially interested companies (eg Italian Society of Anesthesiology)
Increase the sensitivity of doctors and operators on the problems of the elderly population with hip fracture between participating centers | Entire study duration, approximately 5 years
  Increase the sensitivity of doctors and operators participating in the study and of potential other operators belonging to other centers on the problems of the elderly population with hip fracture, ensuring periodic (half-yearly / annual) a return of information (through general reports and by centers) to participating centers explaining the clinical and management characteristics of patients
Enhance the model of orthogeriatrics and geriatric-orthopedic management | Entire study duration, approximately 5 years
  Enhance the model of orthogeriatrics and geriatric-orthopedic management, through analyzes that study the relationship between the model of care received and clinical outcomes (onset of post-operative complications, recovery of the ability to walk, destination for discharge)

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (11):
  - Ospedale S. Agostino Estense, Baggiovara
  - Policlinico S.Orsola-Malpighi, Bologna
  - Ospedale Centrale di Bolzano, Bolzano
  - ASST Vimercate - Ospedale di Carate Brianza, Carate Brianza
  - Arcispedale Sant'Anna, Ferrara
  - A.O.U. di Careggi, Florence
  - Azienda Usl Toscana centro, Florence
  - Ospedale Galliera Genova, Genova
  - Ospedale Policlinico S. Martino, Genova
  - Policlinico Universitario Campus Bio-Medico, Roma
  - ASST della Valtellina e dell'Alto Lario, Sondrio